CLINICAL TRIAL: NCT00050323
Title: Phase 1/2 Study to Assess the Safety and Efficacy of Vaccinations With Allogeneic Dendritic Cells: Autologous Tumor-Derived Cells Subjected to Electrofusion in Patients With AJCC Stage IV Renal Cell Carcinoma
Brief Title: Safety/Efficacy of a Vaccine Prepared From Dendritic Cells Combined With Tumor Cells to Treat Advanced Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCREN-005-01; NCT00062192 (obsolete NCT alias)
Record Dates: First submitted 2002-12-04; First posted 2002-12-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Carcinoma, Renal Cell
Keywords: Stage IV Renal Cell Carcinoma; Kidney Cancer; Cancer (General)
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Neoplasms

INTERVENTIONS:
Drug: Allogeneic DCs and Autologous RCC Tumor Derived Cells

SUMMARY:
The primary purpose of this study is to determine the safety of injections prepared from donor blood cells fused to a patient's own tumor cells which are then used to treat advanced (Stage IV) kidney cancer (renal cell carcinoma or RCC). The study will also explore the effect the injections have on the size of the tumor and the response in the patient's immune system following administration.

DETAILED DESCRIPTION:
Approximately 30,000 new cases of kidney cancer will be diagnosed in the U.S. in 2002, with renal cell carcinoma (RCC) being the most commonly diagnosed type. For patients with locally advanced or metastatic disease, the treatment options are extremely limited and additional options are warranted. Although RCC is generally considered resistant to chemotherapy, spontaneous regressions in patients with metastatic disease have led to research involving immune-mediated therapeutic approaches. Clinical responses have been observed and additional immune-modulating therapeutics are being studied.

Several such approaches have used dendritic cells (DCs), which are known to be potent antigen presenting cells. An antigen is a protein that, when shown to the immune system in the right way, can trigger the cells of the immune system to recognize, remember and eliminate other cells that also display that specific antigen. The cancerous cells in tumors present antigens in such a way that the body's immune system often fails to recognize and eliminate them. It is theorized that when DCs are fused to tumor cells the resulting fused cells will be capable of presenting tumor antigens in an enhanced manner, thus allowing the body's immune system to recognize the tumor antigens on the cancer itself. If this occurs, the patient's immune system may be specifically stimulated, producing a clinically meaningful immune response against the tumor.

In this study DCs produced from healthy volunteer donors (allogeneic DCs) will be fused to the patient's own tumor cells (autologous tumor cells), using an electrical current. The fused dendritic/tumor cells will be returned to the patient in a series of vaccines, six weeks apart.

The purpose of this trial is to determine whether fusing autologous tumor with allogeneic DCs will, with limited associated toxicity, present tumor antigen in such a way as to stimulate an immune response and also show evidence of tumor response.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be greater than or equal to 18 years of age.
* The patient must be diagnosed with AJCC Stage IV (primary or relapsed) Renal Cell Carcinoma.
* The patient must have a Screening Eastern Cooperative Oncology Group (ECOG) Clinical Performance Status of 0-1.
* The patient must have accessible tumor (minimum of 2.5 cm in diameter in aggregate and accessible as defined in the clinical protocol) for vaccine production.
* The patient must have measurable tumor lesions (using Response Evaluation Criteria in Solid Tumors [RECIST]) following resection of tumor lesion(s) used for vaccine production. If the patient has received previous radiation or intra-tumoral investigational treatments, the measurable disease must be outside the previous radiation port or treatment area unless there is documented tumor progression following the completion of therapy.
* The patient must have adequate hematologic, hepatic, and renal function parameters at Screening: White blood cell (WBC) count greater than or equal to 3,000 cells/mm3; Platelet count greater than or equal to 100,000 platelets /mm3; Creatinine (serum) less than 2.0 mg/dL; Total bilirubin less than 2.0 mg/dL; Serum glutamic pyruvate transaminase (SGPT)/alanine aminotransferase (ALT) less than 2.0 x Upper limits of normal; Serum glutamic oxaloacetic transaminase (SGOT)/ aspartate aminotransferase (AST) less than 2.0 x Upper limits of normal
* The patient must be serologically negative for human immunodeficiency virus (HIV)-1, HIV-2, and human T lymphotropic virus (HTLV)-1.
* Female patients of childbearing potential must have negative pregnancy tests, refrain from nursing and must agree to use appropriate contraception for the duration of the trial.
* The patient must have signed and dated written informed consent prior to any study procedures. The consent process must be documented in the patient's medical record.

Exclusion Criteria:

* The patient has received prior chemotherapy for the treatment of RCC.
* The patient has received more than 2 prior regimens for treatment of RCC and the most recent is within 2 weeks of the first screening procedure.
* The patient has received radiation therapy within 2 weeks of the first screening procedure.
* The patient has a clinically significant autoimmune disorder.
* The patient has an active infection at the time of the first screening procedure requiring parenteral antibiotics.
* The patient has clinically significant hematologic, cardiac, renal, or hepatic disease or any other underlying condition that would contraindicate study therapy or confuse interpretation of study results.
* The patient has a history of more than one brain metastasis. Patients with a history of a single brain metastasis must have completed definitive treatment for this metastasis not less than 12 weeks prior to the time of first screening procedure and have remained clinically stable during this interval.
* The patient has a previous unrelated malignancy or second malignancy within 5 years prior to the first screening procedure, except for non-melanoma skin cancer and in situ carcinomas.
* The patient is receiving chronic immunosuppressive and/or oral steroid treatment.
* The patient has any other reason in the Investigator's opinion that would make protocol compliance unmanageable or may compromise the patient's ability to give informed consent.
* The patient has been treated with a non-oncologic investigational drug, biologic or medical device within 30 days of the first screening procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-11; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCLA Medical Center, Los Angeles, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute (DFCI), Boston, Massachusetts
  - The Cleveland Clinic Foundation, Cleveland, Ohio